CLINICAL TRIAL: NCT01251978
Title: Phase 2 Study to Evaluate the Efficacy of High Dose Ranibizumab as Adjuvant in the Treatment of Choroidal Melanoma
Brief Title: Ranibizumab as Adjuvant Therapy for the Treatment of Choroidal Melanoma (Cohort 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New England Retina Associates (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FVF4927s
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Choroidal Melanoma
Keywords: Choroidal melanoma; Ranibizumab; Transpupillary Thermotherapy; CSTIP; Indocyanine Green
MeSH Terms: conditions — Uveal Melanoma | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose Ranibizumab (Active Comparator): 6 patients will receive 3 injections of Ranibizumab (2 mg) a month apart.
  Interventions: Drug: Ranibizumab 2 mg
- Standard Dose Ranibizumab (Active Comparator): 6 patients will receive 0.5 mg of Ranibizumab every two weeks per 3 months.
  Interventions: Drug: 0.5 mg Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab 2 mg — intravitreal injections of ranibizumab once a month, times 3.
  Arms: High dose Ranibizumab
Drug: 0.5 mg Ranibizumab — 6 intravitreal injections of 0.5 mg Ranibizumab every 2 weeks x 3 months.
  Arms: Standard Dose Ranibizumab

SUMMARY:
Ranibizumab has proven to be of benefit to improve the perfusion in the retina of patients with Choroidal Melanoma. The investigators consider that higher doses of Ranibizumab can help reduce the number of laser treatments that might be needed to control the tumor.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Primary pigmented or amelanotic choroidal melanoma measuring 16 mm or less in the largest basal diameter and 6 mm or less in the apical height.
* Location of the tumor, posterior to the equator of the eye.
* Documented growth of tumor by A-B scan.
* Ability to provide written informed consent and comply with the study assessment for the full duration of the study.

Exclusion Criteria:

* Pregnancy or lactation.
* Premenopausal women not using adequate contraception.
* Current infection or inflammation in either eye.
* Extension of tumor into the orbit.
* Regional spread or metastatic disease.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Any known allergy to any of the components to be used in the study.
* Participation in another simultaneous medical investigation or trial.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Liggett, MD, Principal Investigator — New England Retina Associates
Locations (1):
- New England Retina Associates, Hamden, Connecticut, United States

REFERENCES:
- See also: New England Retina Associates website. It contains all the clinical trials that we are running. — http://www.retinamd.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants were enrolled - 2 participants were eliminated early in the study for non compliance.
Groups:
- High Dose Ranibizumab: patients will receive 3 injections of Ranibizumab (2 mg) a month apart.
  Ranibizumab 2 mg: intravitreal injections of ranibizumab once a month, times 3.
- Standard Dose Ranibizumab: patients will receive 0.5 mg of Ranibizumab every two weeks per 3 months.
  0.5 mg Ranibizumab: 6 intravitreal injections of 0.5 mg Ranibizumab every 2 weeks x 3 months.
Period: Overall Study
Arm/Group | High Dose Ranibizumab | Standard Dose Ranibizumab
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Ranibizumab | Standard Dose Ranibizumab | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Safety/Efficacy of Intravitreal Injection of High Dose Ranibizumab Combined With TTT + ICG-based Photodynamic Therapy in the Treatment of Choroidal Melanoma by Reporting the Number of Participants With Complications.
Time Frame: 1 year
Population: complications were only assessed in the high dose group
Measure: Number; unit: participant
Arm/Group | High Dose Ranibizumab
Number analyzed (Participants) | 5
participant
  vascular occlusion | 4
  retinal detachment | 1
  persistent sub retinal fluid (srf) | 1
  CME | 1
  metastatic death | 1

2. Secondary Outcome: Tumor Thickness
Time Frame: baseline and 1 year
Measure: Mean (Full Range); unit: millimeters (mm)
Arm/Group | High Dose Ranibizumab | Standard Dose Ranibizumab
Number analyzed (Participants) | 5 | 3
millimeters (mm)
  baseline | 4.85 [2.5 to 7.48] | 2.91 [2.5 to 3.5]
  12 month | 2.68 [NA to NA] — no measure of dispersion is available - PI left and there is no data available | 0.79 [NA to NA] — no measure of dispersion is available - PI left and there is no data available

3. Secondary Outcome: Visual Acuity (LogMar)
Time Frame: 12 months
Measure: Number; unit: LogMar
Arm/Group | High Dose Ranibizumab | Standard Dose Ranibizumab
Number analyzed (Participants) | 5 | 3
LogMar
  Patient 01 | NA — not applicable for this arm | 0.1
  Patient 02 | NA — not applicable for this arm | 0.1
  Patient 03 | NA — not applicable for this arm | 1.21
  Patient 04 | 2.3 | NA — not applicable for this arm
  Patient 05 | 2.3 | NA — not applicable for this arm
  Patient 06 | 0.1 | NA — not applicable for this arm
  Patient 07 | 0 | NA — not applicable for this arm
  Patient 08 | 1.3 | NA — not applicable for this arm

ADVERSE EVENTS:
Description: Adverse event data are not available to be reported per group or according to severity because the PI left the institution and adverse event data in the required format is not available.
Arm/Group | High Dose Ranibizumab | Standard Dose Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes